CLINICAL TRIAL: NCT05092607
Title: Evaluation of the Detection Performance of the N Antigenemia of SARS-CoV-2 in the General Population for the Diagnosis and Screening of COVID-19
Acronym: CoviBlood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021 A00515 36
Record Dates: First submitted 2021-10-01; First posted 2021-10-25 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Viral Infection
Keywords: COVID-19 diagnostic

STUDY DESIGN:
Intervention Model Description: Cross-sectional study
Masking Description: 267 Symptomatic hospitalized patients 400 Symptomatic or symptomatic patients not hospitalized 800 asymptomatic patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venous and Capillary blood sampling (Experimental): Venous and Capillary blood sampling
  Interventions: Diagnostic Test: Venous and Capillary blood sampling

INTERVENTIONS:
Diagnostic Test: Venous and Capillary blood sampling — Venous sample at the bend of the elbow (7mL) taken immediately after the nasopharyngeal sample.
  Capillary blood sampling, for patients included in participating centers

SUMMARY:
SARS-CoV-2 is responsible for COVID-19. Today, RT-PCR performed on a nasopharyngeal sample remains the gold standard for diagnosing SARS-CoV-2 infection. However, several other assays have been developed to increase testing capabilities and provide rapid screening strategies such as antigenic lateral flow assays. Most recommended tests to date are based nasopharyngeal sampling that is often poorly tolerated by patients and associated with a significant risk of infection for the sampler. Saliva can be used but provide slightly lower sensitivities depending of the subsequent assay use with those samples. The detection of the N antigen of SARS-CoV-2, by ELISA or rapid immunochromatographic technique, on a serum or blood sample would make it possible to overcome these constraints and to provide a new testing alternative. ELISA tests are faster, cheaper and easier to automate than molecular biology approaches.

Blood sampling may be easier to perform in certain populations (in particular in hospitalized patients who already benefit from blood sampling, blood donors, etc.), require less equipment, and is better tolerated (immunocompromised patients subject to blood sampling repeated), and can be integrated more systematically into assessments carried out at the entrance to hospitals or in town, etc. If the N-antigen levels in blood are sufficient, rapid antigen assay on capillary blood could also provide useful testing alternatives.

In a pilot study conducted at Bichat Claude Bernard Hospital, the sensitivity of the first available commercial test was estimated at 93% (95% CI, 84.7-100), and its specificity at 98% (95% CI, 85.3-100).

The main objective of the current work is to evaluate the sensitivity of the SARS-CoV-2 N antigen detection in the serum compared to nasopharyngeal SARS-CoV-2 PCR in several populations such as symptomatic hospitalized patients, symptomatic non-hospitalized patients and asymptomatic subjects.

For each detection kit evaluated, the primary endpoint is the sensitivity (and its 95% confidence interval) of the detection of SARS-CoV-2 N antigen in serum overall and in those populations. The specificity will also be assess.

DETAILED DESCRIPTION:
SARS-CoV-2 is responsible for the COVID-19 pathology. Since the emergence of the virus in China at the end of 2019, the virus has become pandemic and responsible for constant epidemic waves since 2020. France was hit by a first epidemic wave from February to April 2020. This epidemic wave could only be stopped by the implementation of national containment. The virus continues to circulate in France and has been accelerating since the end of August in the general population. The fight against this expansion and new waves aims to slow the viral expansion, to allow the development of new knowledge, treatments and vaccine approaches, as well as to limit the use of intensive care units, so as not to exceed their reception capacities. This fight involves in particular the use of broad and rapid screening practices in the general population in the event of symptoms, events inducing at risk contacts or travel. Today, gold standard assays are the reference methods of RT-PCR on nasopharyngeal swabs. The general population still has great difficulties in finding an available screening center and obtaining a result in a short time, allowing effective isolation and investigation of cases. Alternatives are being used to increase testing capabilities: (i) detection of the N antigen on a nasopharyngeal sample, however with less sensitivity than RT-PCR (ii) saliva sampling but mostly limited, in France, to children population as less sensitive than nasopharyngeal sampling.

Today, only RT-PCR performed on a nasopharyngeal sample therefore remains the reference technique for diagnosing SARS-CoV-2 infection. This method has several flaws, in particular for mass screening. Thus, (i) RT-PCR can only be carried out in laboratories suitable for molecular biology approaches, limiting the number of centers and sometimes imposing significant transport delays; (ii) RT-PCR is a technique requiring long turn around times, rarely compatible with rapid screening strategies; (iii) RT-PCR is relatively expensive; (iv) the nasopharyngeal sample is a sample that is often poorly tolerated by patients and associated with a non-negligible risk of infection for the medical staff performing the sampling. Several other approaches have been evaluated to overcome these difficulties. Antigenic detection of SARS-CoV-2 on nasopharyngeal swab: these approaches were authorized by the French HAS authorities for symptomatic patients. The sensitivity is more limited than with RT-PCR approaches and still potentially infectious viral loads (between 25 and 33 Ct) may not be detected. PCR detection of SARS-CoV-2 on saliva sample allow to avoid the constraints of nasopharyngeal samples but present a sensitivity issue, especially in patients with little or no symptoms. Recently, a new approach, based on the detection of the N antigen of the virus in a blood sample, has been described. The first commercially available method was evaluated at the Virology laboratory at Bichat Hospital in the case of a retrospective study on frozen serum samples. This innovative approach shows satisfactory sensitivity in hospitalized patients. Sensitivity was estimated to be 93.0% (95% CI: 84.7-100) within the first 14 days after symptom onset among 165 patients tested with PCR positive for SARS-CoV-2. The sensitivity was better for high viral loads (49 positives out of 50 with a viral load <30 Ct obtained in the same 24 hours as the serum sample). The specificity, estimated on 63 non-COVID patients, was 98.4% (95% CI: 85.3 to 100). This first study included few outpatients

ELIGIBILITY:
Inclusion Criteria:

* Subject informed and having signed the consent
* Age ≥ 18 years old
* Affiliation to a social security
* Indication for carrying out a screening or diagnostic test for COVID-19

For the study of diagnostic performance in symptomatic hospitalized patients, at least one of the following criteria (HAS recommendations - June 2020):

* Respiratory rate> 25 / min
* Pulse> 100 / mn
* SpO2 <94%
* Dyspnea

For the study of diagnostic performance in asymptomatic patients:

● No symptoms of respiratory infection present (fever, chills, sweating, headache, myalgia, feeling sick, cough, rhinorrhea or sputum, sore throat, chest pain)

For the study of diagnostic performance in symptomatic or pauci-symptomatic patients who are not hospitalized:

● None of the criteria of the two previous populations

Exclusion Criteria:

* Contraindication to performing a nasopharyngeal sample or inability to perform the nasopharyngeal sample
* Subject who has already participated in the study
* All categories of persons protected according to the CSP (minor subject, pregnant, deprived of liberty, under measure of legal protection, guardianship or curators)
* Lack of social security affiliation, CMU (or equivalent)
* Subject under AME
* Lack of signed informed consent

For the study of diagnostic performance in pauci-symptomatic patients

• Need for nasal oxygen therapy

For the study of diagnostic performance in asymptomatic patients

* Presence of respiratory symptoms suggestive of viral infection of the upper respiratory tract
* Need for nasal oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1467 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of the sensitivity of detection of SARS-CoV-2 N antigen | 1 day
  The sensitivity corresponds to the number of patients with a positive detection of SARS-CoV-2 antigenemia and a positive SARS-CoV-2 nasopharyngeal PCR / Number of patients with a positive SARS-CoV-2 nasopharyngeal PCR

CONTACTS AND LOCATIONS:
Overall Officials: VISSEAUX BENOIT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France